CLINICAL TRIAL: NCT02386072
Title: A Prospective, Non-interventional, Registry Study of Patients Initiating a Course of DrugTherapy for Overactive Bladder (OAB)
Brief Title: A Prospective, Observational, Multicenter Study of Patients Following Initiation of a New Course of Treatment for Overactive Bladder (OAB)
Acronym: PERSPECTIVE
Status: Completed | Type: Observational
Sponsor: Astellas Scientific & Medical Affairs, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 178-MA-1006
Record Dates: First submitted 2015-03-06; First posted 2015-03-11 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2018-10

CONDITIONS: Urinary Bladder Overactive; Overactive Bladder; Urinary Bladder Diseases; Urologic Diseases
Keywords: Betanis®; Myrbetriq®; Quality of Life; Antimuscarinics; Betmiga®; Overactive Bladder; Observational
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Bladder Diseases; Urologic Diseases | interventions — mirabegron; Tolterodine Tartrate; oxybutynin; darifenacin; trospium chloride; Solifenacin Succinate; fesoterodine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1. patients diagnosed with OAB taking mirabegron: patients diagnosed with OAB whose physician has decided to prescribe mirabegron as part of routine clinical practice
  Interventions: Drug: mirabegron
- 2. patients diagnosed with OAB taking an antimuscarinic: patients diagnosed with OAB whose physician has decided to prescribe an antimuscarinic as part of routine clinical practice
  Interventions: Drug: antimuscarinic medication

INTERVENTIONS:
Drug: mirabegron — oral
  Other Names: YM178; Betanis; Myrbetriq; Betmiga
  Groups: 1. patients diagnosed with OAB taking mirabegron
Drug: antimuscarinic medication — oral
  Other Names: Ditropan XL; Gelnique; Enablex; Trosec; Sanctura; Oxybutynin IR; Vesicare; Oxytrol; Toviaz; Detrol
  Groups: 2. patients diagnosed with OAB taking an antimuscarinic

SUMMARY:
A study to identify factors that are associated with improved effectiveness in pharmacologic therapy of Overactive Bladder, from the patient perspective primarily measured by OAB-Q-SF (Overactive Bladder Questionnaire Short Form)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with OAB (with or without urgency incontinence) by the treating HCP, with symptoms for at least three months prior to study enrollment
* Initiating a new course of treatment with mirabegron or antimuscarinic medication (including patch formulation) for OAB, which may be first course of any treatment for OAB, restart or switch from one drug to another
* Willing and able to complete PRO questionnaires with minimal assistance

Exclusion Criteria:

* Current participation in clinical trials of OAB
* Use of more than one OAB medication at time of enrollment
* Patients whose OAB has been treated with onabotulinumtoxinA, sacral neuromodulation, percutaneous tibial nerve stimulation, external beam radiation (XRT), stents, surgery, or intermittent catheterization prior to or at time of enrollment
* Neurologic conditions associated with OAB symptoms
* Patients residing in a nursing home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sites that include medical specialties involved in the treatment of OAB, such as general practice/internal medicine, nurse practitioners, obstetricians/ gynecologists, urologists, and uro-gynecologists
Sampling Method: Non-Probability Sample
Enrollment: 1524 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in OAB-related QoL and symptom bother | Baseline, Month 1, 3, 6 and 12
  Overactive Bladder (OAB), Quality of Life (QoL). As measured by the Overactive Bladder Questionnaire Short Form (OAB-Q-SF) questionnaire scores

SECONDARY OUTCOMES:
Effectiveness as measured by impression of severity of OAB | Baseline, Month 1, 3, 6 and 12
  Via the Patient Perception of Bladder Condition [PPBC]
Effectiveness as measured by general health related QoL | Baseline, Month 1, 3, 6 and 12
  via the EuroQol 5D [EQ-5D]
Persistence with OAB drug treatment | Baseline till End of Study (ESV) (up to month 12)
  The duration of time a patient continues to take the prescribed medication
Use of additional (add-on) medications | Baseline till ESV (up to month 12)
  As reported by patients and HCP
Switching of medication | Baseline till ESV (up to month 12)
  As reported by patients and HCP
OAB drug treatment satisfaction | Baseline, month 1, 3, 6 and 12
  Via the Overactive Bladder Treatment Satisfaction Questionnaire (OAB-S)
Reasons for switching of medication | Baseline till ESV (up to month 12)
  As reported by patients and HCP for each specific medication, number and percent
Reasons for discontinuation of medication | Baseline till ESV (up to month 12)
  As reported by patients and HCP for each specific medication, number and percent
Reasons for add-on medication | Baseline till ESV (up to month 12)
  As reported by patients and HCP for each specific medication, number and percent
Reasons for dose titration | Baseline till ESV (up to month 12)
  As reported by patients and HCP for each specific medication
Frequency of dose titration | Baseline till ESV (up to month 12)
  As reported by patients and HCP for each specific medication
Safety profile as assessed by recording AEs and SAEs | Baseline till ESV (up to month 12)
  Adverse Events (AEs), Serious Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Urology, Study Director — Astellas Scientific & Medical Affairs, Inc.
Locations (92):
- United States (75):
  - Site US1051, Birmingham, Alabama
  - Site US1094, Birmingham, Alabama
  - Site US1010, Huntsville, Alabama
  - Site US1020, Mobile, Alabama
  - Site US1006, Goodyear, Arizona
  - Site US1036, Mesa, Arizona
  - Site US1028, Phoenix, Arizona
  - Site US1100, Tucson, Arizona
  - Site US1083, Tucson, Arizona
  - Site US1114, Little Rock, Arkansas
  - Site US1061, Little Rock, Arkansas
  - Site US1112, Garden Grove, California
  - Site US1104, Sacramento, California
  - Site US1013, Santa Ana, California
  - Site US1090, Northglenn, Colorado
  - Site US1050, Hialeah, Florida
  - Site US1068, Miami, Florida
  - Site US1079, Miami, Florida
  - Site US1031, Miami, Florida
  - Site US1032, Miami, Florida
  - Site US1044, Miami, Florida
  - Site US1018, Miami, Florida
  - Site US1098, Miami, Florida
  - Site US1075, Miami, Florida
  - Site US1048, North Miami Beach, Florida
  - Site US1093, Ocoee, Florida
  - Site US1055, Pompano Beach, Florida
  - Site US1042, Atlanta, Georgia
  - Site US1035, Columbus, Georgia
  - Site US1009, Marietta, Georgia
  - Site US1016, Idaho Falls, Idaho
  - Site US1046, Lake Barrington, Illinois
  - Site US1019, Evansville, Indiana
  - Site US1034, Evansville, Indiana
  - Site US1097, Muncie, Indiana
  - Site US1017, Council Bluffs, Iowa
  - Site US1064, Overland Park, Kansas
  - Site US1077, Lafayette, Louisiana
  - Site US1058, Annapolis, Maryland
  - Site US1088, Burlington, Massachusetts
  - Site US1059, Fall River, Massachusetts
  - Site US1076, Watertown, Massachusetts
  - Site US1089, Worcester, Massachusetts
  - Site US1062, Hamtramck, Michigan
  - Site US1047, Hazelwood, Missouri
  - Site US1082, St Louis, Missouri
  - Site US1105, St Louis, Missouri
  - Site US1102, Omaha, Nebraska
  - Site US1039, Omaha, Nebraska
  - Site US1043, Las Vegas, Nevada
  - Site US1052, Las Vegas, Nevada
  - Site US1085, New Brunswick, New Jersey
  - Site US1001, Sicklerville, New Jersey
  - Site US1008, Albuquerque, New Mexico
  - Site US1103, Buffalo, New York
  - Site US1096, Garden City, New York
  - Site US1106, New York, New York
  - Site US1111, New York, New York
  - Site US1040, Newburgh, New York
  - Site US1045, Poughkeepsie, New York
  - Site US1060, Raleigh, North Carolina
  - Site US1007, Hilliard, Ohio
  - Site US1021, Downingtown, Pennsylvania
  - Site US1070, Providence, Rhode Island
  - Site US1004, Myrtle Beach, South Carolina
  - Site US1084, Sioux Falls, South Dakota
  - Site US1015, Clarksville, Tennessee
  - Site US1037, Fort Worth, Texas
  - Site US1080, Houston, Texas
  - Site US1067, Houston, Texas
  - Site US1057, Katy, Texas
  - Site US1012, Plano, Texas
  - Site US1099, Virginia Beach, Virginia
  - Site US1086, Seattle, Washington
  - Site US1071, Monroe, Wisconsin
- Canada (17):
  - Site CA1026, Calgary, Alberta
  - Site CA1066, Coquitlam, British Columbia
  - Site CA1000, Victoria, British Columbia
  - Site CA1022, Burlington, Ontario
  - Site CA1029, Burlington, Ontario
  - Site CA1005, Greater Sudbury, Ontario
  - Site CA1072, Kingston, Ontario
  - Site CA1023, London, Ontario
  - Site CA1014, Mississauga, Ontario
  - Site CA1095, Oshawa, Ontario
  - Site CA1025, Oshawa, Ontario
  - Site CA1065, Ottawa, Ontario
  - Site CA1101, Richmond Hill, Ontario
  - Site CA1054, Scarborough Village, Ontario
  - Site CA1027, Toronto, Ontario
  - Site CA1092, Toronto, Ontario
  - Site CA1038, Pointe-Claire, Quebec

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Carlson KV, Rovner ES, Nair KV, Deal AS, Kristy RM, Schermer CR. Factors Associated with Improvements in Patient-Reported Outcomes During Mirabegron or Antimuscarinic Treatment of Overactive Bladder Syndrome: A Registry Study (PERSPECTIVE). Adv Ther. 2019 Aug;36(8):1906-1921. doi: 10.1007/s12325-019-00994-7. Epub 2019 Jun 20. PMID 31222714
- [Derived] Rovner ES, Carlson KV, Deal AS, Nair KV, Oakkar EE, Park J, Gemmen E, Kristy RM, Gooch KL, Schermer CR. A Prospective, non-intErventional Registry Study of PatiEnts initiating a Course of drug Therapy for overactIVE bladder (PERSPECTIVE): Rationale, design, and methodology. Contemp Clin Trials. 2018 Jul;70:83-87. doi: 10.1016/j.cct.2018.05.006. Epub 2018 May 16. PMID 29777865